CLINICAL TRIAL: NCT00006009
Title: A Phase I, Multiple Dose Escalation Trial of Intravenous Humanized Anti-CD3 Antibody (HuM291) in Patients With CD3+ T-cell Lymphomas
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Advanced or Recurrent Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SUMC-NCI-102; CDR0000068017 (Registry Identifier: PDQ (Physician Data Query)); NCI-102
Record Dates: First submitted 2000-07-05; First posted 2003-10-08 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2003-04

CONDITIONS: Lymphoma; Small Intestine Cancer
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome | interventions — visilizumab

INTERVENTIONS:
Biological: visilizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have advanced or recurrent lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of monoclonal antibody HuM291 in patients with advanced or recurrent CD3+ T-cell lymphomas.
* Evaluate the pharmacokinetics and pharmacodynamics of this treatment regimen in this patient population.
* Determine the response in these patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive monoclonal antibody HuM291 IV over 3 hours on days 1-4 in the absence of unacceptable toxicity. Patients achieving a partial response, complete response with recurrence, or stable disease may receive further therapy.

Cohorts of 3-6 patients receive escalating doses of monoclonal antibody HuM291 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed weekly for 1 month and then monthly for 3 months.

PROJECTED ACCRUAL: A total of 12-15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD3+ T-cell lymphoma for which no standard curative therapy exists

  * Peripheral T-cell lymphoma

    * Recurrent and/or progressive disease after at least 1 prior therapy
  * Mycosis fungoides

    * Stage IB/IIA

      * Recurrent and/or progressive disease after at least 2 prior therapies
    * Stage IIB-IVB

      * Recurrent and/or progressive disease after at least 1 prior therapy
  * All other T-cell lymphomas

    * Recurrent and/or progressive disease after at least 1 prior therapy
* Evaluable disease

  * Any nodal site or mass lesion at least 1.5 cm in longest axis on physical exam or CT scan
  * Skin lesions at least 1 cm in longest axis for cutaneous lymphoma
* High numbers of circulating T-cells allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2
* Karnofsky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm^3*
* Absolute neutrophil count at least 1,000/mm^3*
* Platelet count at least 75,000/mm^3* NOTE: * Unless due to lymphoma

Hepatic:

* Bilirubin no greater than 2.0 times normal*
* AST/ALT no greater than 2.5 times upper limit of normal*
* Hepatitis B and C negative NOTE: * Unless due to lymphoma

Renal:

* Not specified

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No other uncontrolled illness
* No ongoing or active infection
* No other active malignancies except basal cell skin cancer or carcinoma in situ of the cervix
* HIV-1 negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Biologic therapy:

* At least 60 days since prior humanized or chimeric antibody therapy

Chemotherapy:

* At least 3 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 30 days since prior investigational drugs or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youn H. Kim, MD, Study Chair — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States